CLINICAL TRIAL: NCT05150067
Title: Efficacy of a Blended Learning Programme in Enhancing the Communication Skill Competence and Self-Efficacy of Nursing Students in Conducting Clinical Handovers: A Randomised Controlled Trial
Brief Title: A Blended Learning to Enhance Communication Skill Competence and Self-Efficacy of Nursing Students in Clinical Handovers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Ho Cheung William, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 19-622
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2021-12

CONDITIONS: Self Efficacy; Nursing; Communication
Keywords: Blended learning; online module; clinical handover; communication skill competence; self-efficacy; nursing students
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor was blinded to the group assignment so that the scores remained unbiased.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The participants in the experimental group received a blended learning programme with face-to-face training and an online module on handover practice.
  Interventions: Other: A Blended Learning Programme
- waitlist control group (Active Comparator): The participants in the waitlist control group received the same face-to-face training workshop as the experimental group. However, these participants were invited to access the online module only after data collection was completed.
  Interventions: Other: Waitlist control group

INTERVENTIONS:
Other: A Blended Learning Programme — A blended learning programme with face-to-face training and an online module on handover practice
  Arms: Experimental group
Other: Waitlist control group — The participants in the waitlist control group received the same face-to-face training workshop as the experimental group. However, these participants were invited to access the online module only after data collection was completed
  Arms: waitlist control group

SUMMARY:
This study aimed to examine the efficacy of a blended learning programme in enhancing the communication skill competence and self-efficacy of final-year nursing students in conducting clinical handovers.

DETAILED DESCRIPTION:
A clinical handover refers to the process of transferring the relevant information and facilitating continuity of patient care from one healthcare provider to another. It is an essential nursing practice that ensures patient safety. The information transmitted during the handover must be clear, concise and systematic to facilitate the provision of continuous patient care. Ambiguous communication and unsystematically transmitted information can often impede the clarity of ideas, result in the omission of important patient information and delay medical treatment, consequently endangering the safety of patients. Nursing students and newly graduated nurses often struggle with clinical handovers due to a lack of communication skill competence and self-efficacy in performing this practice.

Blended learning programmes (BLPs) are commonly used as constructivist pedagogical approaches in nursing education. BLPs have been used successfully to teach theoretical courses and psychomotor skills in nursing education and have been proven to benefit the knowledge, self-efficacy, motivation, attitudes and perceived competence of students. However, no studies that examine the efficiency of BLPs in enhancing the communication skill competence and self-efficacy of nursing students in conducting clinical handovers have been found. Therefore, this study aimed to determine the efficacy of BLP in improving the communication skill competence and self-efficacy of nursing students in conducting clinical handovers.

ELIGIBILITY:
Inclusion Criteria:

* were Hong Kong residents who could speak Cantonese and read Chinese and English
* were aged at least 18 years
* had not previously enrolled in a clinical handover training programme.

Exclusion Criteria:

- NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline communication skill competence at 2 weeks after they received the intervention | From baseline to 2 weeks after they received the intervention
  The participants' communication skill competence in conducting clinical handovers was assessed using the Situation, Background, Assessment, Recommendation (SBAR) Communication and Communication Clarity tool. The assessment had 23 items that were rated on a Likert scale. Higher scores correspond to better performance.

SECONDARY OUTCOMES:
Change from baseline self-perceived communication self-efficacy level in conducting clinical handovers at 2 weeks after they received the intervention | From baseline to 2 weeks after they received the intervention
  The participants' self-perceived communication self-efficacy level in conducting clinical handovers was assessed using a visual analogue scale. The visual analogue scale values were found to reliably reflect the participants' true attitudes with low distortion and bias. The participants were requested to drag a sliding bar from 0 to 100 on the online survey platform to indicate the level of confidence in their ability to conduct clinical handovers (0 = Not at all confident, 100 = Extremely confident).

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Study Director — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung JYS, Li WHC, Cheung AT, Ho LLK, Chung JOK. Efficacy of a blended learning programme in enhancing the communication skill competence and self-efficacy of nursing students in conducting clinical handovers: a randomised controlled trial. BMC Med Educ. 2022 Apr 13;22(1):275. doi: 10.1186/s12909-022-03361-3. PMID 35418214